CLINICAL TRIAL: NCT02273765
Title: Phase III Open-label Randomized Multicenter Trial to Assess the Non-inferiority of Raltegravir Compared With EFavirenz, Both in Combination With LAmivudine and TEnofovir, in ART-naïve HIV-1-infected Patients Receiving Rifampin for Active TuBerculosis
Brief Title: Raltegravir Versus Efavirenz in Naive HIV-1-infected Patients Receiving Rifampin for Active Tuberculosis
Acronym: REFLATE TB2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry); Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12300 REFLATE TB2
Record Dates: First submitted 2014-10-20; First posted 2014-10-24 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: HIV-1 Infection; Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Tenofovir; Lamivudine; Raltegravir Potassium; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir (Active Comparator): Tenofovir 300mg QD + lamivudine 300mg QD + raltegravir 400mg BID
  Interventions: Drug: Tenofovir + lamivudine + raltegravir
- Efavirenz (Experimental): Tenofovir 300mg QD + lamivudine 300mg QD + efavirenz 600mg QD
  Interventions: Drug: Tenofovir + lamivudine + efavirenz

INTERVENTIONS:
Drug: Tenofovir + lamivudine + raltegravir — In this arm, patients will receive the following medications :
  * Tenofovir disoproxil fumarate (TDF) 300 mg / Lamivudine (3TC) 300 mg FDC once a day (1 tablet qd)
  * Raltegravir (RAL) 400 mg (Isentress®): twice daily (1 tablet bid), with food
  In countries where TDF/3TC FDC is not available, the following separate drugs will be used:
  * Tenofovir disoproxil fumarate (TDF) 300 mg (Viread® 245 mg): once a day (1 tablet qd)
  * Lamivudine (3TC) : 300 mg once a day (300 mg, 1 tablet qd or 150 mg 2 tablets qd)
  * Raltegravir (RAL) 400 mg (Insentress®): twice daily (1 tablet bid), with food
  Arms: Raltegravir
Drug: Tenofovir + lamivudine + efavirenz — In this arm, patients will receive the following medications, in accordance with treatment guidelines in all countries:
  * Tenofovir disoproxil fumarate (TDF) 300 mg / lamivudine (3TC) 300 mg FDC once a day (1 tablet qd)
  * Efavirenz (EFV) 600 mg: once a day, at night (1 tablet qd)
  OR:
  • Tenofovir disoproxil fumarate (TDF) 245 300 mg / lamivudine (3TC) 300 mg / efavirenz (EFV) 600 mg: once a day (1 tablet qd), at night, if possible without food
  In countries where TDF/3TC FDC is not available, the following separate drugs will be used:
  * Tenofovir disoproxil fumarate (TDF) 300 mg (Viread® 245 mg): once a day (1 tablet qd)
  * Lamivudine (3TC): 300 mg once a day (300 mg, 1 tablet qd or 150 mg 2 tablets qd)
  * Efavirenz (EFV) 600 mg: once a day, at night (1 tablet qd), if possible without food. The dose will not be adapted to the patient's body weight.
  Arms: Efavirenz

SUMMARY:
Phase III trial evaluating raltegravir as an alternative to efavirenz for antiretroviral treatment of HIV-infected patients with tuberculosis.

DETAILED DESCRIPTION:
Phase III multicenter, international, open-label, randomized trial evaluating non-inferiority of raltegravir at dose of 400mg BID compared to efavirenz 600mg QD, both in association with tenofovir disoproxil fumarate and lamivudine in ART-naïve HIV-1 infected patients with active TB disease receiving a rifampin-based TB treatment initiated <8 weeks before inclusion. Patients will be randomized between 2 arms: the raltegravir (RAL) 400 mg bid arm or the efavirenz (EFV) 600 mg qd arm, each in combination with tenofovir disoproxil fumarate (TDF) and lamivudine (3TC) and will be followed for 48 weeks after entry in the trial (ART initiation).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Aged 18 years or more
* Confirmed HIV-1 infection as documented at any time prior to trial entry per national HIV testing procedures
* ART naïve
* For women of childbearing potential i.e. women of childbearing age who are not menopausal, or permanently sterilized (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy) or not refraining from sexual activity: negative urinary test for pregnancy and acceptance to use contraceptive methods
* Confirmed or probable active TB disease of any location, except neurological (meningitis or encephalitis), according to the following criteria based on WHO updated definitions:

  * Bacteriologically confirmed pulmonary TB (PTB) or extrapulmonary TB (EPTB), e.g. TB with a biological specimen positive by smear microscopy, culture or nucleic acid amplification test (such as Xpert MTB/RIF).
  * Clinically diagnosed PTB or EPTB with typical histological evidence of TB (caseous or granulomatous) on biopsy specimen or positive urinary LAM test OR a significant improvement on TB treatment
* Ongoing standard rifampin-containing TB treatment for ≤8 weeks at inclusion
* For French patients, affiliation to a Social Security program

Exclusion Criteria:

* HIV-2 co-infection
* Impaired hepatic function (icterus or ALT (SGPT) > 5ULN)
* Hemoglobin < 6.5 g/dl
* Creatinine clearance <60ml/min (assessed by the Cockroft and Gault formula)
* Mycobacterium tuberculosis strain resistant to rifampin (current or past history).
* Neurological TB (meningitis or encephalitis)
* Severe associated diseases requiring specific treatment (including all specific AIDS defining illnesses other than TB, and any severe sepsis)
* Any condition which might, in the investigator's opinion, compromise the safety of treatment and/or patient's adherence to trial procedures including very severe TB-related clinical condition
* Concomitant treatments including phenytoin or phenobarbital (compounds interacting with UGT1A1)
* For HCV co-infected patients, need to start specific treatment for hepatitis during the trial duration
* For women of childbearing potential:

  * Pregnancy or breastfeeding
  * Refusal to use a contraceptive method
  * Any history of ARV intake for prevention of mother to child transmission of HIV (pMTCT)
* Subjects participating in another clinical trial evaluating therapies and including an exclusion period that is still in force during the screening phase
* Person under guardianship, or deprived of freedom by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in virologic success | Week 48
  Virologic success, defined as plasma HIV-1 RNA <50 copies/mL, at week 48 with a window period of 42 to 54 weeks (snapshot algorithm). Discontinuation of the strategy (ie. permanent discontinuation of EFV, RAL), missing values, loss to follow-up and death will be considered as failure.

SECONDARY OUTCOMES:
Time to death | Week 48
Frequency, type and time to new or recurrent AIDS-defining illnesses | Week 48
Frequency, type and time to severe HIV-associated non-AIDS defining illnesses | Week 48
Frequency, type and time to grade 3 or 4 adverse events | Week 48
Frequency, type and time to drug-induced clinical or biological adverse reactions of grade 3 or 4 or leading to treatment interruption | Week 48
Change in plasma HIV-1 RNA from baseline to week 48 | Week 48
Proportion of patients in virologic success at each time point (HIV-1 RNA<50 copies/mL) | Week 48
Time to virologic failure during follow-up | Week 48
Frequency and time to new antiretroviral genotypic resistance in plasma RNA in patients with virologic failure | Week 48
Change in CD4 cell counts from baseline to week 48 | Week 48
Frequency, type and time to Immune Reconstitution Inflammatory Syndrome | Week 48
Frequency of tuberculosis treatment outcomes | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Grinsztejn, MD, PhD, Study Chair — Laboratory on Clinical research on DST/AIDS-IPEC FIOCRUZ Av Brasil, 4365 Manguinhos Rio de Janeiro, Brazil CEP 21040-900; Nathalie De Castro, MD, Study Chair — AP-HP Hôpital Saint-Louis 1 avenue Claude Vellefaux, 75010 Paris, France
Locations (5):
- Laboratory of clinical research on STD/AIDS - IPEC/FIOCRUZ, Rio de Janeiro, Brazil
- PACCI / CePReF Centre de Prise en charge de Recherche et de Formation, Abidjan, Côte d’Ivoire
- Hôpital Saint Louis, Paris, France
- Instituto Nacional de Saude / Hospital Geral de Machava, Maputo, Mozambique
- Pham Ngoc Thach Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] De Castro N, Marcy O, Chazallon C, Messou E, Eholie S, N'takpe JB, Bhatt N, Khosa C, Timana Massango I, Laureillard D, Chau GD, Domergue A, Veloso V, Escada R, Wagner Cardoso S, Delaugerre C, Anglaret X, Molina JM, Grinsztejn B; ANRS 12300 Reflate TB2 study group. Standard dose raltegravir or efavirenz-based antiretroviral treatment for patients co-infected with HIV and tuberculosis (ANRS 12 300 Reflate TB 2): an open-label, non-inferiority, randomised, phase 3 trial. Lancet Infect Dis. 2021 Jun;21(6):813-822. doi: 10.1016/S1473-3099(20)30869-0. Epub 2021 Mar 2. PMID 33667406